CLINICAL TRIAL: NCT00105157
Title: Multicenter Study to Evaluate the Safety and Efficacy of MK0518 in Combination With An Optimized Background Therapy (OBT), Versus OBT Alone, in HIV-Infected Patients With Documented Resistance
Brief Title: Safety and Efficacy of an Investigational Drug in Human Immunodeficiency Virus (HIV)-Infected Patients Failing Current Antiretroviral Therapies (0518-005)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0518-005; MK0518-005; 2005_007
Record Dates: First submitted 2005-03-08; First posted 2005-03-09 (Estimated); Results first posted 2010-04-12 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: HIV Infections; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Raltegravir Potassium

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1 (Experimental): MK0518 200 mg
  Interventions: Drug: Comparator: MK0518
- 2 (Experimental): MK0518 400 mg
  Interventions: Drug: MK0518
- 3 (Experimental): MK0518 600 mg
  Interventions: Drug: MK0518
- 4 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Comparator: MK0518 — MK0518 oral tablets 200 mg b.i.d, for 24 weeks
  Other Names: MK0518
  Arms: 1
Drug: MK0518 — MK0518 oral tablets 400 mg b.i.d, for 24 weeks
  Arms: 2
Drug: MK0518 — MK0518 oral tablets 600 mg b.i.d, for 24 weeks
  Arms: 3
Drug: Placebo — Placebo to MK0518, oral tablet b.i.d, for 24 weeks
  Arms: 4

SUMMARY:
This study will investigate the safety and efficacy of different doses of an investigational drug (MK0518) as a therapy for HIV-infected patients failing current antiretroviral therapies.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be HIV positive with Human Immunodeficiency Virus (HIV) Ribonucleic Acid (RNA) values that are within ranges required by the study
* Patient must be currently on antiretroviral therapy (ART)

Exclusion Criteria:

* Patient less than 18 years of age
* Additional exclusion criteria will be discussed and identified by the study doctor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2005-03; Primary Completion 2006-10 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Grinsztejn B, Nguyen BY, Katlama C, Gatell JM, Lazzarin A, Vittecoq D, Gonzalez CJ, Chen J, Harvey CM, Isaacs RD; Protocol 005 Team. Safety and efficacy of the HIV-1 integrase inhibitor raltegravir (MK-0518) in treatment-experienced patients with multidrug-resistant virus: a phase II randomised controlled trial. Lancet. 2007 Apr 14;369(9569):1261-1269. doi: 10.1016/S0140-6736(07)60597-2. PMID 17434401

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Primary therapy period: 22-Apr-2005 to 09-Nov-2006
  Multicenter (31) in the United States (15) and outside the United States (16)
Pre-assignment Details: Patients failed prior antiretroviral therapy (HIV RNA >5000 copies/mL), and had documented resistance to at least one drug in each class of licensed oral antiretroviral therapy (Nucleoside Reverse Transcriptase inhibitors, Non-Nucleoside Reverse Transcriptase inhibitors and Protease Inhibitors). All patients must have met laboratory criteria.
Groups:
- MK0518 200 mg b.i.d.: Optimized background antiretroviral therapy (OBT), if possible, based on screening genotypic/phenotypic resistance and past treatment history and MK0518 200 mg twice a day (b.i.d.). Once the Phase III dose was determined, all patients were switched to the Phase III dose (400 mg b.i.d.) after completion of at least 24 weeks double-blind therapy.
- MK0518 400 mg b.i.d.: OBT, if possible, based on screening genotypic/phenotypic resistance and past treatment history and MK0518 400 mg b.i.d.
- MK0518 600 mg b.i.d.: OBT, if possible, based on screening genotypic/phenotypic resistance and past treatment history and MK0518 600 mg b.i.d.. Once the Phase III dose was determined, all patients were switched to the Phase III dose (400 mg b.i.d.) after completion of at least 24 weeks double-blind therapy.
- Placebo: OBT, if possible, based on screening genotypic/phenotypic resistance and past treatment history and MK0518 matching placebo b.i.d.. Once the Phase III dose was determined, all patients were switched to the Phase III dose (400 mg b.i.d.) after completion of at least 24 weeks double-blind therapy.
Period: Double-Blind (DB)
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Started | 44 | 45 | 45 | 45
Treated | 43 | 45 | 45 | 45
Completed | 30 | 31 | 33 | 6
Not Completed | 14 | 14 | 12 | 39
Not completed — Never Treated | 1 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 1 | 1
Not completed — Lack of Efficacy | 11 | 14 | 11 | 38
Period: Open-Label Continuation of DB
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Started | 30 | 31 | 33 | 6
Completed | 23 | 21 | 24 | 5
Not Completed | 7 | 10 | 9 | 1
Not completed — Adverse Event | 3 | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 4 | 3 | 1
Not completed — Lost to Follow-up | 1 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 3 | 0
Not completed — Patient did not continue in extension | 1 | 0 | 0 | 0
Not completed — Patient moved/site stopped trial | 1 | 3 | 2 | 0
Period: Open-Label Post Virologic Failure(OLPVF)
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Started | 11 (Number of Patients appropriate for and who consented to enter the OLPVF) | 13 (Number of Patients appropriate for and who consented to enter the OLPVF) | 11 (Number of Patients appropriate for and who consented to enter the OLPVF) | 37 (Number of Patients appropriate for and who consented to enter the OLPVF)
Completed | 2 | 7 | 5 | 19
Not Completed | 9 | 6 | 6 | 18
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 7 | 6 | 5 | 10
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 5
Not completed — Patient moved/Site stopped trial | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo | Total
Number analyzed (Participants) | 43 | 45 | 45 | 45 | 178
Age, Continuous [Mean (Full Range); unit: years] | 44.0 [18 to 57] | 45.1 [32 to 69] | 43.8 [25 to 63] | 43.3 [29 to 59] | 44.1 [18 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 4 | 5 | 21
  Male | 36 | 40 | 41 | 40 | 157
Race/Ethnicity, Customized [Number; unit: participants]
  White | 36 | 35 | 32 | 33 | 136
  Black | 3 | 5 | 7 | 5 | 20
  Asian | 0 | 0 | 2 | 1 | 3
  Hispanic | 4 | 5 | 4 | 5 | 18
  Others | 0 | 0 | 0 | 1 | 1
Cluster of Differentiation 4 (CD4) Cell Count [Mean (Full Range); unit: Cells/mm3] | 244.9 [30 to 1153] | 220.6 [68 to 673] | 220.4 [30 to 663] | 274.0 [37 to 880] | 239.9 [30 to 1153]
Plasma HIV RNA [Mean (Full Range); unit: log10 copies/mL] | 4.6 [3.5 to 5.9] | 4.8 [3.7 to 5.9] | 4.7 [3.8 to 5.8] | 4.7 [3.6 to 5.8] | 4.7 [3.5 to 5.9]
Plasma Human Immunodeficiency Virus (HIV) Ribonucleic Acid (RNA) [Mean (Full Range); unit: Copies/mL] | 44642.6 [3000 to 750000] | 59107.9 [4770 to 750000] | 49064.8 [7030 to 589000] | 47432.6 [3630 to 611000] | 49841.6 [3000 to 750000]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Plasma HIV RNA (log10 Copies/mL) at Week 24
Description: Mean change from baseline at Week 24 in HIV RNA (log10 copies/mL) in all patients
Time Frame: Baseline and Week 24
Population: Observed mean change from baseline in log10 Plasma HIV RNA for each group was calculated using the conventional imputation (replace HIV RNA <400 copies/mL by 400 copies/mL if signal detected, or 200 copies/mL if signal not detected). Missing values: baseline-carry-forward for all failures or discontinued due to lack of efficacy
Measure: Mean (95% Confidence Interval); unit: HIV RNA (log10 copies/mL)
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 43 | 45 | 45 | 45
HIV RNA (log10 copies/mL) | -1.80 [-2.10 to -1.50] | -1.87 [-2.16 to -1.58] | -1.84 [-2.10 to -1.58] | -0.35 [-0.61 to -0.09]

2. Secondary Outcome: Number of Patients With Virologic Responses at Week 24
Description: Number of patients who achieve HIV RNA <400 copies/mL; HIV RNA level <50 copies/mL at Week 24; or reduction from baseline in HIV RNA (log10 copies/mL) exceeding 1.0 log10 copies/mL at Week 24; at Week 24
Time Frame: 24 weeks
Population: All patients who took study medication and had HIV RNA tests performed were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 43 | 45 | 45 | 45
Participants
  HIV RNA <400 copies/mL | 30 | 32 | 32 | 7
  HIV RNA <50 copies/mL | 28 | 25 | 30 | 6
  >1.0 log10 Drop in HIV RNA | 33 | 36 | 36 | 8

3. Secondary Outcome: Change From Baseline in CD4 Cell Count at Week 24
Description: Mean change from baseline at Week 24 in CD4 Cell Count (cells/mm3)
Time Frame: Baseline and Week 24
Population: Observed failure approach assuming baseline-carry-forward for all failures, exclude other missing values. Baseline CD4 Cell Count (cells/mm3) was carried forward for patients who discontinued assigned therapy due to lack of efficacy.
Measure: Mean (95% Confidence Interval); unit: CD4 Cell Count (cells/mm3)
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 43 | 45 | 45 | 45
CD4 Cell Count (cells/mm3) | 62.9 [27.8 to 97.9] | 112.8 [75.7 to 150.0] | 94.1 [60.1 to 128.0] | 5.4 [-9.9 to 20.7]

4. Secondary Outcome: Number of Patients With Clinical Adverse Experiences (CAEs) at 48 Weeks
Description: An adverse experience (AE) is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR'S product, whether or not considered related to the use of the product
Time Frame: 48 weeks
Population: All patients who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 43 | 45 | 45 | 45
Participants
  With CAEs | 37 | 37 | 41 | 37
  Without CAEs | 6 | 8 | 4 | 8

5. Secondary Outcome: Number of Patients With Serious CAEs at 48 Weeks
Description: Serious CAEs are any AEs occurring at any dose that; Results in death; or Is life threatening; or Results in a persistent or significant disability/incapacity; or Results in or prolongs an existing inpatient hospitalization; or Is a congenital anomaly/birth defect; or Is a cancer; or Is an overdose
Time Frame: 48 weeks
Population: All patients who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 43 | 45 | 45 | 45
Participants
  With Serious CAEs | 3 | 7 | 4 | 3
  Without Serious CAEs | 40 | 38 | 41 | 42

6. Secondary Outcome: Number of Patients With Drug-related CAEs at 48 Weeks
Description: Patients with drug-related (as assessed by an investigator who is a qualified physician according to his/her best clinical judgment) CAEs
Time Frame: 48 weeks
Population: All patients who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 43 | 45 | 45 | 45
Participants
  With Drug-Related CAEs | 18 | 19 | 24 | 24
  Without Drug-Related CAEs | 25 | 26 | 21 | 21

7. Secondary Outcome: Number of Patients With Serious Drug-related CAEs at 48 Weeks
Description: Serious CAEs are any AEs occurring at any dose that; Results in death; or Is life threatening; or Results in a persistent or significant disability/incapacity; or Results in or prolongs an existing inpatient hospitalization; or Is a congenital anomaly/birth defect; or Is a cancer; or Is an overdose. Drug-related are as assessed by an investigator who is a qualified physician according to his/her best clinical judgment.
Time Frame: 48 weeks
Population: All patients who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 43 | 45 | 45 | 45
Participants
  With Serious Drug-Related CAEs | 1 | 0 | 1 | 2
  Without Serious Drug-Related CAEs | 42 | 45 | 44 | 43

8. Secondary Outcome: Number of Patients That Died by 48 Weeks
Time Frame: 48 weeks
Population: All patients who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 43 | 45 | 45 | 45
Participants
  Died | 1 | 0 | 1 | 0
  Did not Die | 42 | 45 | 44 | 45

9. Secondary Outcome: Number of Patients That Discontinued With CAEs at 48 Weeks
Time Frame: 48 weeks
Population: All patients who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 43 | 45 | 45 | 45
Participants
  Discontinued With CAEs | 1 | 0 | 1 | 1
  Did Not Discontinue With CAEs | 42 | 45 | 44 | 44

10. Secondary Outcome: Number of Patients That Discontinued With Drug-related CAEs at 48 Weeks
Time Frame: 48 weeks
Population: All patients who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 43 | 45 | 45 | 45
Participants
  Discontinued With Drug-related CAEs | 0 | 0 | 0 | 1
  Did Not Discontinue With Drug-related CAEs | 43 | 45 | 45 | 44

11. Secondary Outcome: Number of Patients That Discontinued With Serious CAEs at 48 Weeks
Time Frame: 48 weeks
Population: All patients who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 43 | 45 | 45 | 45
Participants
  Discontinued With Serious CAEs | 1 | 0 | 1 | 1
  Did Not Discontinue With Serious CAEs | 42 | 45 | 44 | 44

12. Secondary Outcome: Number of Patients That Discontinued With Serious Drug-related CAEs at 48 Weeks
Time Frame: 48 weeks
Population: All patients who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 43 | 45 | 45 | 45
Participants
  Discontinued With Serious Drug-related CAEs | 0 | 0 | 0 | 1
  Did Not Discontinue With Serious Drug-related CAEs | 43 | 45 | 45 | 44

13. Secondary Outcome: Number of Patients With Laboratory Adverse Experiences (LAEs) at 48 Weeks
Description: A laboratory adverse experience (LAE) is defined as any unfavorable and unintended change in the chemistry of the body temporally associated with the use of the SPONSOR'S product, whether or not considered related to the use of the product
Time Frame: 48 weeks
Population: All patients who took study medication and had any laboratory tests performed were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 43 | 45 | 45 | 45
Participants
  With LAEs | 10 | 12 | 14 | 11
  Without LAEs | 33 | 33 | 31 | 34

14. Secondary Outcome: Number of Patients With Drug-related LAEs at 48 Weeks
Description: Patients with drug-related (as assessed by an investigator who is a qualified physician according to his/her best clinical judgment) LAEs
Time Frame: 48 weeks
Population: All patients who took study medication and had any laboratory tests performed were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 43 | 45 | 45 | 45
Participants
  With Drug-related LAEs | 7 | 8 | 7 | 8
  Without Drug-related LAEs | 36 | 37 | 38 | 37

15. Secondary Outcome: Number of Patients Discontinued With Laboratory Adverse Experiences (LAEs) at 48 Weeks
Time Frame: 48 weeks
Population: All patients who took study medication and had any laboratory tests performed were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 43 | 45 | 45 | 45
Participants
  Discontinued With LAEs | 1 | 0 | 0 | 0
  Did Not Discontinue With LAEs | 42 | 45 | 45 | 45

16. Secondary Outcome: Number of Patients Discontinued With Drug-related LAEs at 48 Weeks
Time Frame: 48 weeks
Population: All patients who took study medication and had any laboratory tests performed were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 43 | 45 | 45 | 45
Participants
  Discontinued With Drug-Related LAEs | 1 | 0 | 0 | 0
  Did Not Discontinue With Drug-Related LAEs | 42 | 45 | 45 | 45

17. Secondary Outcome: Number of Patients With Clinical Adverse Experiences (CAEs) at 96 Weeks
Description: as for outcome 4
Time Frame: 96 weeks
Population: All patients who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 43 | 45 | 45 | 45
Participants
  With CAEs | 43 | 42 | 45 | 38
  Without CAEs | 0 | 3 | 0 | 7

18. Secondary Outcome: Number of Patients With Serious CAEs at 96 Weeks
Description: as for outcome 5
Time Frame: 96 weeks
Population: All patients who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 43 | 45 | 45 | 45
Participants
  With Serious CAEs | 4 | 9 | 5 | 3
  Without Serious CAEs | 39 | 36 | 40 | 42

19. Secondary Outcome: Number of Patients With Drug-related CAEs at 96 Weeks
Description: as for outcome 6
Time Frame: 96 weeks
Population: All patients who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 43 | 45 | 45 | 45
Participants
  With drug-related CAEs | 24 | 25 | 28 | 26
  Without drug-related CAEs | 19 | 20 | 17 | 19

20. Secondary Outcome: Number of Patients With Serious Drug-related CAEs at 96 Weeks
Description: as for outcome 7
Time Frame: 96 weeks
Population: All patients who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 43 | 45 | 45 | 45
Participants
  With Serious Drug-Related CAEs | 1 | 0 | 1 | 2
  Without Serious Drug-Related CAEs | 42 | 45 | 44 | 43

21. Secondary Outcome: Number of Patients That Died by 96 Weeks
Time Frame: 96 weeks
Population: All patients who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 43 | 45 | 45 | 45
Participants
  Died | 2 | 1 | 1 | 0
  Did Not Die | 41 | 44 | 44 | 45

22. Secondary Outcome: Number of Patients That Discontinued With CAEs at 96 Weeks
Time Frame: 96 weeks
Population: All patients who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 43 | 45 | 45 | 45
Participants
  Discontinued With CAEs | 2 | 1 | 1 | 1
  Did Not Discontinue With CAEs | 41 | 44 | 44 | 44

23. Secondary Outcome: Number of Patients That Discontinued With Drug-related CAEs at 96 Weeks
Time Frame: 96 weeks
Population: All patients who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 43 | 45 | 45 | 45
Participants
  Discontinued With Drug-Related CAEs | 0 | 0 | 0 | 1
  Did Not Discontinue With Drug-Related CAEs | 43 | 45 | 45 | 44

24. Secondary Outcome: Number of Patients That Discontinued With Serious CAEs at 96 Weeks
Time Frame: 96 weeks
Population: All patients who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 43 | 45 | 45 | 45
Participants
  Discontinued With Serious CAEs | 2 | 1 | 1 | 1
  Did Not Discontinue With Serious CAEs | 41 | 44 | 44 | 44

25. Secondary Outcome: Number of Patients That Discontinued With Serious Drug-related CAEs at 96 Weeks
Time Frame: 96 weeks
Population: All patients who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 43 | 45 | 45 | 45
Participants
  Discontinued With Serious Drug-related CAEs | 0 | 0 | 0 | 1
  Did Not Discontinue With Serious Drug-related CAEs | 43 | 45 | 45 | 44

26. Secondary Outcome: Number of Patients With Laboratory Adverse Experiences (LAEs) at 96 Weeks
Description: as for outcome 13
Time Frame: 96 weeks
Population: All patients who took study medication and had any laboratory tests performed were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 43 | 45 | 45 | 45
Participants
  With LAEs | 12 | 15 | 17 | 12
  Without LAEs | 31 | 30 | 28 | 33

27. Secondary Outcome: Number of Patients With Drug-related LAEs at 96 Weeks
Description: as for outcome 14
Time Frame: 96 weeks
Measure: Number; unit: Participants
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 43 | 45 | 45 | 45
Participants
  With Drug-Related LAEs | 9 | 9 | 11 | 8
  Without Drug-Related LAEs | 34 | 36 | 34 | 37

28. Secondary Outcome: Number of Patients Discontinued With Laboratory Adverse Experiences (LAEs) at 96 Weeks
Time Frame: 96 weeks
Population: All patients who took study medication and had any laboratory tests performed were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 43 | 45 | 45 | 45
Participants
  Discontinued With LAEs | 1 | 1 | 0 | 0
  Did Not Discontinue With LAEs | 42 | 44 | 45 | 45

29. Secondary Outcome: Number of Patients Discontinued With Drug-related LAEs at 96 Weeks
Time Frame: 96 weeks
Population: All patients who took study medication and had
  any laboratory tests performed were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 43 | 45 | 45 | 45
Participants
  Discontinued With Drug-related LAEs | 1 | 1 | 0 | 0
  Did Not Discontinue With Drug-related LAEs | 42 | 44 | 45 | 45

30. Post Hoc Outcome: Number of Patients With Virologic Responses at Week 168 in Combined Substudies
Description: Number of patients who achieve HIV RNA <400 copies/mL; HIV RNA level <50 copies/mL at Week 168; or reduction from baseline in HIV RNA (log10 copies/mL) exceeding 1.0 log10 copies/mL at Week 168.
Time Frame: 168 weeks
Population: Analysis population is based on the modified intent to treat (MITT) approach, where patients are included in the treatment group to which they were randomized. Patients who were randomized but never dosed are not included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 43 | 43 | 44 | 45
Participants
  HIV RNA <400 copies/mL | 21 | 15 | 22 | 5
  HIV RNA <50 copies/mL | 20 | 13 | 19 | 5
  >1.0 log10 Drop in HIV RNA | 22 | 15 | 23 | 5

31. Other Pre Specified Outcome: Change From Baseline in Plasma HIV RNA (log10 Copies/mL) at Week 168 in Combined Substudies
Description: Mean change from baseline at Week 168 in HIV RNA (log10 copies/mL) in patients from combined substudies in the double-blind plus open-label phases.
Time Frame: Baseline and Week 168
Population: as for outcome 30
Measure: Mean (95% Confidence Interval); unit: HIV RNA (log10 copies/mL)
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 37 | 38 | 40 | 44
HIV RNA (log10 copies/mL) | -1.67 [-2.17 to -1.18] | -1.32 [-1.88 to -0.77] | -1.66 [-2.15 to -1.17] | -0.33 [-0.61 to -0.04]

32. Other Pre Specified Outcome: Change From Baseline in CD4 Cell Count at Week 168 in Combined Substudies
Description: Mean change from baseline at Week 168 in CD4 Cell Count (cells/mm3) in patients from combined substudies in the double-blind plus open-label phases.
Time Frame: Baseline and Week 168
Population: as for outcome 30
Measure: Mean (95% Confidence Interval); unit: CD4 Cell Count (cells/mm3)
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 36 | 38 | 39 | 44
CD4 Cell Count (cells/mm3) | 96.9 [58.7 to 135.1] | 107.7 [49.4 to 165.9] | 147.4 [86.5 to 208.3] | 25.5 [-1.1 to 52.0]

33. Secondary Outcome: Number of Patients With Clinical Adverse Experiences (CAEs) at 168 Weeks
Description: as for outcome 4
Time Frame: 168 weeks
Population: All patients who took study medication were included in the analysis (All Patients as Treated approach). Data include patients from the double-blind plus open-label phases.
Measure: Number; unit: Participants
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 43 | 45 | 45 | 45
Participants
  With CAEs | 43 | 43 | 45 | 38
  Without CAEs | 0 | 2 | 0 | 7

34. Secondary Outcome: Number of Patients With Serious CAEs at 168 Weeks
Description: as for outcome 5
Time Frame: 168 weeks
Population: as for outcome 33
Measure: Number; unit: Participants
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 43 | 45 | 45 | 45
Participants
  With Serious CAEs | 6 | 13 | 7 | 3
  Without Serious CAEs | 37 | 32 | 38 | 42

35. Secondary Outcome: Number of Patients With Drug-related CAEs at 168 Weeks
Description: as for outcome 6
Time Frame: 168 weeks
Population: as for outcome 33
Measure: Number; unit: Participants
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 43 | 45 | 45 | 45
Participants
  With Drug-Related CAEs | 27 | 27 | 30 | 26
  Without Drug-Related CAEs | 16 | 18 | 15 | 19

36. Secondary Outcome: Number of Patients With Serious Drug-related CAEs at 168 Weeks
Description: as for outcome 7
Time Frame: 168 weeks
Population: as for outcome 33
Measure: Number; unit: Participants
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 43 | 45 | 45 | 45
Participants
  With Serious Drug-Related CAEs | 2 | 0 | 2 | 2
  Without Serious Drug-Related CAEs | 41 | 45 | 43 | 43

37. Secondary Outcome: Number of Patients That Died by 168 Weeks
Time Frame: 168 weeks
Population: as for outcome 33
Measure: Number; unit: Participants
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 43 | 45 | 45 | 45
Participants
  Died | 3 | 1 | 1 | 0
  Did not Die | 40 | 44 | 44 | 45

38. Secondary Outcome: Number of Patients That Discontinued With CAEs at 168 Weeks
Time Frame: 168 weeks
Population: as for outcome 33
Measure: Number; unit: Participants
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 43 | 45 | 45 | 45
Participants
  Discontinued With CAEs | 3 | 1 | 1 | 1
  Did Not Discontinue With CAEs | 40 | 44 | 44 | 44

39. Secondary Outcome: Number of Patients That Discontinued With Drug-related CAEs at 168 Weeks
Time Frame: 168 weeks
Population: as for outcome 33
Measure: Number; unit: Participants
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 43 | 45 | 45 | 45
Participants
  Discontinued With Drug-related CAEs | 0 | 0 | 0 | 1
  Did Not Discontinue With Drug-related CAEs | 43 | 45 | 45 | 44

40. Secondary Outcome: Number of Patients That Discontinued With Serious CAEs at 168 Weeks
Time Frame: 168 weeks
Population: as for outcome 33
Measure: Number; unit: Participants
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 43 | 45 | 45 | 45
Participants
  Discontinued With Serious CAEs | 3 | 1 | 1 | 1
  Did Not Discontinue With Serious CAEs | 40 | 44 | 44 | 44

41. Secondary Outcome: Number of Patients That Discontinued With Serious Drug-related CAEs at 168 Weeks
Time Frame: 168 weeks
Population: as for outcome 33
Measure: Number; unit: Participants
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 43 | 45 | 45 | 45
Participants
  Discontinued With Serious Drug-related CAEs | 0 | 0 | 0 | 1
  Did Not Discontinue With Serious Drug-related CAEs | 43 | 45 | 45 | 44

42. Secondary Outcome: Number of Patients With Laboratory Adverse Experiences (LAEs) at 168 Weeks
Description: as for outcome 13
Time Frame: 168 weeks
Population: as for outcome 33
Measure: Number; unit: Participants
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 43 | 45 | 45 | 45
Participants
  With LAEs | 17 | 16 | 18 | 12
  Without LAEs | 26 | 29 | 27 | 33

43. Secondary Outcome: Number of Patients With Serious LAEs at 168 Weeks
Description: Serious LAEs are any LAEs occurring at any dose that; Results in death; or Is life threatening; or Results in a persistent or significant disability/incapacity; or Results in or prolongs an existing inpatient hospitalization; or Is a congenital anomaly/birth defect; or Is a cancer; or Is an overdose
Time Frame: 168 weeks
Population: as for outcome 33
Measure: Number; unit: Participants
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 43 | 45 | 45 | 45
Participants
  With Serious LAEs | 1 | 0 | 1 | 0
  Without Serious LAEs | 42 | 45 | 44 | 45

44. Secondary Outcome: Number of Patients Discontinued With Drug-related LAEs at 168 Weeks
Time Frame: 168 weeks
Population: as for outcome 33
Measure: Number; unit: Participants
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 43 | 45 | 45 | 45
Participants
  Discontinued With Drug-Related LAEs | 2 | 0 | 0 | 0
  Did Not Discontinue With Drug-Related LAEs | 41 | 45 | 45 | 45

45. Secondary Outcome: Number of Patients With Drug-related LAEs at 168 Weeks
Description: as for outcome 14
Time Frame: 168 weeks
Population: as for outcome 33
Measure: Number; unit: Participants
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 43 | 45 | 45 | 45
Participants
  With Drug-related LAEs | 13 | 10 | 11 | 9
  Without Drug-related LAEs | 30 | 35 | 34 | 36

46. Secondary Outcome: Number of Patients With Serious Drug-related LAEs at 168 Weeks
Description: as for outcome 43
Time Frame: 168 weeks
Population: as for outcome 33
Measure: Number; unit: Participants
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 43 | 45 | 45 | 45
Participants
  With Drug-related LAEs | 1 | 0 | 1 | 0
  Without Drug-related LAEs | 42 | 45 | 44 | 45

47. Secondary Outcome: Number of Patients Discontinued With LAEs at 168 Weeks
Time Frame: 168 weeks
Population: as for outcome 33
Measure: Number; unit: Participants
Arm/Group | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 43 | 45 | 45 | 45
Participants
  Discontinued With LAEs | 2 | 0 | 0 | 0
  Did Not Discontinue With LAEs | 41 | 45 | 45 | 45

ADVERSE EVENTS:
Time Frame: 168 weeks: Due to a 3:1 randomization of MK0518 to placebo and more discontinuations for placebo in the double-blind phase, exposure for MK0518 and placebo differs significantly with follow-up times of 336.3 and 39.7 patient-years, respectively.
Description: AEs were assessed by the investigators.
Groups:
- MK0518: Includes patients from the MK0518 200 mg, 400 mg, and 600 mg b.i.d. dose groups. Patients who completed at least 24 weeks of double-blind therapy without virologic failure entered the open-label phase to receive open-label MK0518 400 mg b.i.d.
Arm/Group | MK0518 | Placebo
Serious Adverse Events (participants affected / at risk) | 28/133 | 3/45
Other Adverse Events (participants affected / at risk) | 131/133 | 39/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MK0518 (N=133) | Placebo (N=45)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0
Atrioventricular Block Complete (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Cardio-Respiratory Arrest (Cardiac disorders) | 1 | 0
Coronary Artery Disease (Cardiac disorders) | 2 | 0
Myocardial Infarction (Cardiac disorders) | 2 | 0
Photophobia (Eye disorders) | 1 | 0
Anogenital Dysplasia (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Irritable Bowel Syndrome (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 1 | 0
Varices Oesophageal (Gastrointestinal disorders) | 1 | 0
Oedema Peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 0
Bile Duct Obstruction (Hepatobiliary disorders) | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Portal Hypertension (Hepatobiliary disorders) | 1 | 0
Anogenital Warts (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Herpes Simplex (Infections and infestations) | 1 | 0
Herpes Zoster (Infections and infestations) | 1 | 0
Leishmaniasis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Postoperative Wound Infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Splenic Abscess (Infections and infestations) | 1 | 0
Staphylococcal Abscess (Infections and infestations) | 1 | 0
Staphylococcal Infection (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 0 | 1
Accidental Overdose (Injury, poisoning and procedural complications) | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Lipase Increased (Investigations) | 1 | 0
Platelet Count Decreased (Investigations) | 1 | 0
Metabolic Acidosis (Metabolism and nutrition disorders) | 1 | 0
Anal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anal Cancer Stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hodgkin's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Facial Palsy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 1
Lacunar Infarction (Nervous system disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 2 | 0
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lipoatrophy (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Shock (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MK0518 (N=133) | Placebo (N=45)
Anaemia (Blood and lymphatic system disorders) | 3 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 11 | 2
Splenomegaly (Blood and lymphatic system disorders) | 3 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Cardiovascular Disorder (Cardiac disorders) | 0 | 1
Cerumen Impaction (Ear and labyrinth disorders) | 3 | 0
Ocular Icterus (Eye disorders) | 3 | 0
Vision Blurred (Eye disorders) | 1 | 1
Abdominal Discomfort (Gastrointestinal disorders) | 4 | 1
Abdominal Distension (Gastrointestinal disorders) | 4 | 1
Abdominal Pain (Gastrointestinal disorders) | 13 | 4
Abdominal Pain Upper (Gastrointestinal disorders) | 5 | 1
Anal Fissure (Gastrointestinal disorders) | 1 | 1
Anogenital Dysplasia (Gastrointestinal disorders) | 2 | 1
Cheilitis (Gastrointestinal disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 6 | 1
Diarrhoea (Gastrointestinal disorders) | 29 | 11
Dry Mouth (Gastrointestinal disorders) | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 5
Flatulence (Gastrointestinal disorders) | 3 | 2
Gastric Disorder (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 3 | 1
Hypoaesthesia Oral (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 21 | 10
Periodontitis (Gastrointestinal disorders) | 0 | 1
Tongue Ulceration (Gastrointestinal disorders) | 4 | 0
Toothache (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 11 | 2
Asthenia (General disorders) | 6 | 3
Chest Discomfort (General disorders) | 3 | 0
Chest Pain (General disorders) | 4 | 3
Chills (General disorders) | 2 | 1
Drug Intolerance (General disorders) | 0 | 1
Fatigue (General disorders) | 14 | 4
Injection Site Inflammation (General disorders) | 0 | 1
Injection Site Nodule (General disorders) | 3 | 1
Injection Site Reaction (General disorders) | 12 | 3
Nodule (General disorders) | 3 | 0
Oedema Peripheral (General disorders) | 7 | 0
Pain (General disorders) | 4 | 2
Pyrexia (General disorders) | 12 | 1
Sensation Of Pressure (General disorders) | 0 | 1
Hepatic Steatosis (Hepatobiliary disorders) | 4 | 0
Hepatosplenomegaly (Hepatobiliary disorders) | 3 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 | 0
Jaundice (Hepatobiliary disorders) | 3 | 0
Drug Hypersensitivity (Immune system disorders) | 1 | 1
Hypersensitivity (Immune system disorders) | 2 | 1
Acute Tonsillitis (Infections and infestations) | 0 | 1
Anogenital Warts (Infections and infestations) | 7 | 0
Bronchitis (Infections and infestations) | 15 | 7
Candidiasis (Infections and infestations) | 4 | 0
Cellulitis (Infections and infestations) | 3 | 0
Ear Infection (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 3 | 0
Folliculitis (Infections and infestations) | 1 | 1
Fungal Skin Infection (Infections and infestations) | 1 | 2
Furuncle (Infections and infestations) | 3 | 1
Gastroenteritis (Infections and infestations) | 4 | 1
Genital Herpes (Infections and infestations) | 3 | 0
Giardiasis (Infections and infestations) | 0 | 1
Herpes Simplex (Infections and infestations) | 3 | 0
Herpes Virus Infection (Infections and infestations) | 4 | 0
Herpes Zoster (Infections and infestations) | 7 | 1
Influenza (Infections and infestations) | 17 | 2
Nasopharyngitis (Infections and infestations) | 17 | 2
Onychomycosis (Infections and infestations) | 4 | 2
Oral Candidiasis (Infections and infestations) | 5 | 0
Oral Herpes (Infections and infestations) | 2 | 2
Papilloma Viral Infection (Infections and infestations) | 2 | 1
Pharyngitis (Infections and infestations) | 3 | 0
Pharyngotonsillitis (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 3 | 0
Respiratory Tract Infection (Infections and infestations) | 5 | 2
Sinusitis (Infections and infestations) | 7 | 1
Sinusitis Bacterial (Infections and infestations) | 3 | 0
Skin Infection (Infections and infestations) | 1 | 1
Syphilis (Infections and infestations) | 4 | 0
Tooth Abscess (Infections and infestations) | 5 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 13 | 4
Urinary Tract Infection (Infections and infestations) | 4 | 0
Contusion (Injury, poisoning and procedural complications) | 3 | 0
Excoriation (Injury, poisoning and procedural complications) | 3 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 3 | 0
Tibia Fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 8 | 0
Aspartate Aminotransferase Increased (Investigations) | 9 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 3 | 0
Blood Amylase Increased (Investigations) | 6 | 0
Blood Bilirubin Increased (Investigations) | 14 | 2
Blood Cholesterol Increased (Investigations) | 4 | 4
Blood Creatine Phosphokinase Increased (Investigations) | 14 | 0
Blood Creatinine Increased (Investigations) | 4 | 1
Blood Glucose Increased (Investigations) | 6 | 0
Blood Phosphorus Decreased (Investigations) | 2 | 2
Blood Potassium Decreased (Investigations) | 3 | 0
Blood Testosterone Decreased (Investigations) | 1 | 1
Blood Triglycerides Increased (Investigations) | 6 | 2
Blood Urine Present (Investigations) | 3 | 2
Lipase Increased (Investigations) | 7 | 0
Low Density Lipoprotein Increased (Investigations) | 4 | 2
Lymphocyte Count Decreased (Investigations) | 0 | 1
Neutrophil Count Decreased (Investigations) | 4 | 2
Platelet Count Decreased (Investigations) | 3 | 0
Protein Urine Present (Investigations) | 5 | 1
Weight Decreased (Investigations) | 0 | 1
White Blood Cell Count Decreased (Investigations) | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 4 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 3 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 6 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 10 | 1
Muscle Hypertrophy (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 4 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 7 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 10 | 2
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Dizziness (Nervous system disorders) | 5 | 0
Dysgeusia (Nervous system disorders) | 4 | 1
Dysphasia (Nervous system disorders) | 0 | 1
Facial Palsy (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 21 | 5
Hemicephalalgia (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 3 | 1
Migraine (Nervous system disorders) | 0 | 1
Neuropathy Peripheral (Nervous system disorders) | 5 | 2
Paraesthesia (Nervous system disorders) | 8 | 0
Syncope (Nervous system disorders) | 2 | 1
Anxiety (Psychiatric disorders) | 4 | 2
Depression (Psychiatric disorders) | 10 | 1
Insomnia (Psychiatric disorders) | 12 | 2
Sleep Disorder (Psychiatric disorders) | 2 | 1
Dysuria (Renal and urinary disorders) | 3 | 2
Nephrolithiasis (Renal and urinary disorders) | 2 | 1
Renal Cyst (Renal and urinary disorders) | 0 | 1
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 | 1
Erectile Dysfunction (Reproductive system and breast disorders) | 5 | 0
Pelvic Pain (Reproductive system and breast disorders) | 1 | 1
Prostatitis (Reproductive system and breast disorders) | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 23 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Paranasal Sinus Hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 1
Dyshidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 4 | 1
Erythema (Skin and subcutaneous tissue disorders) | 4 | 0
Facial Wasting (Skin and subcutaneous tissue disorders) | 4 | 0
Lipodystrophy Acquired (Skin and subcutaneous tissue disorders) | 6 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 2 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 1
Rash (Skin and subcutaneous tissue disorders) | 9 | 1
Rash Macular (Skin and subcutaneous tissue disorders) | 1 | 1
Rash Papular (Skin and subcutaneous tissue disorders) | 3 | 0
Seborrhoeic Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Lesion (Skin and subcutaneous tissue disorders) | 3 | 0
Skin Nodule (Skin and subcutaneous tissue disorders) | 2 | 1
Subcutaneous Nodule (Skin and subcutaneous tissue disorders) | 4 | 1
Hyperaemia (Vascular disorders) | 3 | 0
Hypertension (Vascular disorders) | 13 | 0

LIMITATIONS AND CAVEATS:
Due to a 3:1 randomization of MK-0518 to placebo and more discontinuations for placebo in the doubleblind phase, exposure for MK-0518 and placebo differs significantly with follow-up times of 336.3 and 39.7 patient-years, respectively.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.